CLINICAL TRIAL: NCT01714310
Title: Characterization and Sequential Pharmacotherapy of Severe Mood Dysregulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Shire (Industry)
Responsible Party: Principal Investigator, James McGough, Professor of Clinical Psychiatry, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U01MH093582 (NIH); U01MH093582 (NIH)
Record Dates: First submitted 2012-10-20; First posted 2012-10-25 (Estimated); Results first posted 2018-02-26 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-01

CONDITIONS: Severe Mood Dysregulation
Keywords: severe mood dysregulation; irritability; lisdexamfetamine; fluoxetine; newly recognized syndrome
MeSH Terms: interventions — Lisdexamfetamine Dimesylate; Fluoxetine

STUDY DESIGN:
Intervention Model Description: Initial arm for open-label titration of lisdexamfetamine followed by randomization of participants who retain eligibility to double blind adjunctive fluoxetine or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Adjunctive fluoxetine (Experimental): Participants previously titrated with open-label lisdexamfetamine randomized to adjunctive fluoxetine at end of study week 4.
  Interventions: Drug: lisdexamfetamine; Drug: fluoxetine
- Adjunctive placebo (Placebo Comparator): Participants previously titrated with open-label lisdexamfetamine randomized to adjunctive placebo at end of study week 4.
  Interventions: Drug: lisdexamfetamine; Drug: Placebo
- Open Lisdexamfetamine Titration (Other): All participants initially titrated with open-label lisdexamfetamine from baseline to end of study week 4.
  Interventions: Drug: lisdexamfetamine

INTERVENTIONS:
Drug: lisdexamfetamine — Titration and open label treatment from baseline visit for 12 week study.
  Other Names: Vyvanse
Drug: Placebo — Initiated at end of study week 4 and continued to study week 12.
  Arms: Adjunctive placebo
Drug: fluoxetine — Initiated at end of study week 4 and continued to study week 12.
  Other Names: Prozac
  Arms: Adjunctive fluoxetine

SUMMARY:
This project will characterize children and adolescents with severe mood dysregulation (SMD) and conduct a pilot study of combination pharmacotherapy as a basis for future intervention trials.

Eligible participants assessed for SMD will have 4 weeks open titration with lisdexamfetamine (LDX) to optimal dose, followed by double-blind randomization to fluoxetine (N=25) or placebo (N=25) in combination with optimized LDX for an additional 8 weeks. Participants will be monitored for clinical response and adverse events.

Specific aims are:

#1: To define youth meeting SMD criteria in terms of psychiatric comorbidity, neurocognitive functioning, and a potential "bio-signature" derived from electroencephalography (EEG).

Specific hypotheses to be tested include: 1) that SMD participants will differ in comparison to non-SMD individuals in our pre-existing database on patterns of a) psychiatric comorbidity, b) symptoms, c) behavioral ratings, and d) neurocognitive functioning, and 2) that a distinct EEG bio-signature will be confirmed in individuals formally diagnosed with SMD.

#2: To conduct a preliminary study of sequential pharmacotherapy for SMD with a stimulant followed by randomized, placebo-controlled selective serotonin re-uptake inhibitor (SSRI) therapy to evaluate the feasibility of recruitment and enrollment and assess the suitability of the proposed combination treatment as a basis for future clinical investigations.

Specific hypotheses to be tested include: 1) that significant improvement in Clinical Global Impression - Improvement -SMD (CGI-I-SMD) scores and other secondary measures are evident after open-label LDX titration; 2) that participants randomized to fluoxetine will demonstrate additional significant improvement in CGI-I-SMD scores and other secondary measures in comparison to participants randomized to placebo; 3) that combination LDX and SSRI therapy is safe and well tolerated, and 4) that EEG profiles will normalize with treatment.

DETAILED DESCRIPTION:
Background

The increased frequency of diagnosed pediatric bipolar disorder has emerged as one of the greatest controversies in child and adolescent psychiatry. Beginning with reports that 20% of prepubertal of children with Attention-Deficit/Hyperactivity Disorder (ADHD) met criteria for juvenile mania, a view arose that bipolar children were more irritable than euphoric and more chronic than episodic, compared with the typical adult. Concurrently, there was a 4 to 6-fold increase in inpatient discharges and 40-fold increase in office-based visits for pediatric bipolar disorder, although many of these failed to meet formal Diagnostic and Statistical Manual (DSM) criteria. Concerns have been raised that any child with impulsive, volatile behavior is apt to be diagnosed as bipolar.

Some attempted to inform valid symptomatic boundaries by proposing a differentiation of narrow versus broad pediatric bipolar phenotypes. The narrow phenotype was defined by strict DSM criteria for mania or hypomania, including discrete episodes of grandiosity and euphoria. In contrast, the broad phenotype, also referred to as severe mood dysregulation (SMD), was defined by chronic, non-episodic illness lacking hallmark symptoms of grandiosity and euphoria, but typified by severe irritability and hyperarousal. Work at the National Institute of Mental Health (NIMH) demonstrated that patterns of adolescent irritability are stable and distinct, with episodic irritability leading to mania and simple phobia, and chronic irritability leading to diagnosed depression and ADHD. On structured assessment, children with SMD were highly comorbid for major depression (20%), anxiety (64%), oppositional defiant disorder (83%), and ADHD (87%). Others also found increased rates of ADHD and anxiety. In addition, the broad and narrow phenotypes could be differentiated according to electroencephalography (EEG) measures. SMD youth have impaired face emotion recognition deficits correlated with dysfunctional family relationships and were less influenced by emotional distracters during tasks of attention. A recent study revealed patterns of amygdala hypoactivation similar to depression, further supporting links between chronic irritability and subsequent depressive episodes.

In response to the perceived over-diagnosis of pediatric DSM bipolar disorder, acknowledgment that the "classic" adult bipolar phenotype does occur in prepubertal youth, and increased recognition that SMD is a distinct behavioral and/or biological syndrome, the DSM-5 Child Disorders Workgroup proposed a new diagnostic category named temper dysregulation disorder with dysphoria (TDD). Criteria for TDD were largely based on SMD, however, the requirement for hyperarousal was removed and minor changes were made in age of onset and exclusion criteria. Unlike SMD, TDD lacks any demonstrated scientific basis or history of prior research. As such, it seems prudent at this time to continue research on the better-established SMD category with an expectation that any information derived will have ready applicability as work on TDD progresses.

One preliminary report suggests that SMD has a lifetime prevalence of 3.3% among those ages 9-19. Recent longitudinal studies further indicate that children with SMD have increased rates of adult mood and anxiety disorders, substance abuse, suicidality, and poorer overall functioning. Given this significant morbidity, it is essential that the investigators increase understanding of children with chronic irritability and affective instability. Impulsive aggression in childhood has been identified as a significant public health concern that cuts across currently defined diagnostic categories. These youth demonstrate increased difficulties with school adjustment, peer interactions, cognitive deficits, problem-solving, and physical abuse - a developmental trajectory predictive of significant adult dysfunction.

Current community practice emphasizes use of second-generation antipsychotic agents for children with impulsive aggression. While risperidone has proven effective for irritability associated with pervasive developmental disorders [25,26] and second-generation antipsychotics have been effective in pediatric bipolar disorder, these agents are associated with significant weight gain and other metabolic effects. Use of these medications is associated with decreased utilization of psychosocial interventions. Given the relationship of SMD with ADHD, anxiety, and unipolar depression, investigations of drugs from other classes with targeted effects and better side effect profiles, such as mood stabilizers, antidepressants, and stimulants, are certainly warranted. In fact, the DSM-5 Workgroup has specifically called for clinical trials stating it is "critically important" to assess whether stimulants and SSRIs should be first line treatments in SMD-affected youth. The only published medication trial in SMD youth is a double-blind placebo controlled study of lithium conducted by the intramural group at NIMH, which failed to demonstrate effects. Other informative investigations include small positive studies of methylphenidate versus placebo for ADHD plus oppositional defiant disorder and aggression, open-label stimulant followed by adjuvant divalproex vs. placebo for ADHD and aggression, and stimulant augmentation with double-blind risperidone versus placebo in ADHD with treatment resistant aggression. These studies are notably heterogeneous in design and choice of outcome measures. No clear predictors of response have been reported.

Most existing SMD research has been conducted by a single intramural group at NIMH. It is imperative that investigations of SMD be expanded to other research groups to ensure that results generalize to broad clinical settings. Additional research is required to delineate clinical phenomenology that will inform subsequent efforts at diagnostic classification. Further work is also necessary to establish the appropriate foundation for future clinical interventions research. This should include pilot studies of various medication classes that might prove useful in management of SMD, as well as examination of various outcome measures that are likely to be useful in both medication and psychosocial intervention trials.

Overview

The study will include comprehensive phenotyping of 65 patients meeting criteria for SMD, including assessment of comorbid psychopathology, language disorder, neurocognition, and EEG. Potential endophenotypes and diagnostic boundaries will be assessed in relation to our large existing database of children and adolescents with internalizing and externalizing disorders, as well as non-clinical controls. Eligible participants with SMD will proceed to a pilot study of sequential pharmacotherapy with an initial 4-week titration of open label lisdexamfetamine (LDX) followed by 8 weeks adjunctive therapy with randomized fluoxetine or placebo. Statistical analyses will address diagnostic boundaries of SMD compared with other disorders and emphasize initial determinations of the potential efficacy and tolerability of stimulant and SSRI treatments for SMD. There will be an added emphasis on effect size estimates and determination of optimal outcome measures in anticipation of future large-scale studies.

Project Visits and Procedures

Following baseline visit (week 0), eligible participants will undergo undergo open-label stepwise titration with one week each of low, medium, and high dose LDX during study weeks 1, 2, and 3. The study physician may modify titration due to emergent side effects following routine practice standards.

At the end of study week 3, the clinician will determine "optimal" stimulant dose based on review of parent and teacher-completed Conners Global Index scales and all available adverse event and side effects data, using procedures similar to those used in other studies. Participants will remain on this optimal stimulant dose for the remainder of the study, unless side effects necessitate some downward dose adjustment.

At study week 4, participants who fail to achieve CGI-I-SMD score < 4 will be randomized to double blind adjunctive treatment with either fluoxetine or placebo.

A forced dose, stepwise, upward titration of one week each of 5, 10, and 20 mg fluoxetine/placebo will occur at during week 5, 6, and 7. The treating physician may modify this titration schedule in response to emergent side effect following routine practice standards. Participants will remain on their week 7 doses of fluoxetine/placebo until the study's final visit, unless side effects necessitate some downward titration.

Side effects, adverse events, and medication compliance will be assessed at each visit. Major outcome assessments will occur at baseline (week 0) , end of week 4, and end of week 12.

Arrangements will be made to transfer participants to standard clinical care following week 12.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants, ages 7-17 years.
2. Abnormal mood (specifically anger, sadness, and/or irritability), present at least half of the day most days and of sufficient severity to be noticeable in the child's environment (e.g. parents, teachers, peers).
3. Hyperarousal, as defined by at least three of the following symptoms: insomnia, agitation, distractibility, racing thoughts or flight of ideas, pressured speech, intrusiveness.
4. Compared to his/her peers, the child exhibits markedly increased reactivity to negative emotional stimuli that is manifest verbally and/or behaviorally. For example, the child responds to frustration with extended temper tantrums (inappropriate for age and/or precipitating event), verbal rages, and/or aggression toward people or property. Such events occur, on average, at least three times a week.
5. Criteria 2, 3, and 4 are currently present and have been present for at least 12 months without any symptom free periods exceeding two months.
6. The onset of symptoms must be prior to age 12 years.
7. The symptoms are severe in at least one setting (e.g. violent outbursts, extreme verbal abuse, assaultiveness at home, school, or with peers). In addition. There are at least mild symptoms (distractibility, intrusiveness) in a second setting.
8. Score > 9 on either the Inattentive or Hyperactive/Impulsive subscales of the baseline ADHD-RS.
9. Score < 12 on the irritability subscale of the Aberrant Behavior Checklist. -

Exclusion Criteria:

1. As evidenced in the mania section of the Kiddie-Schedule for Affective Disorders and Schizophrenia, the individual exhibits any of these cardinal bipolar symptoms in distinct periods lasting more than 1 day, and therefore meets criteria for bipolar disorder not otherwise specified (NOS):

   i) Elevated or expansive mood. ii) Grandiosity or inflated self esteem. iii) Decreased need for sleep. iv) Increase in goal-directed activity (this can result in the excessive involvement in pleasurable activities that have a high potential for painful consequences).
2. Meets criteria for schizophrenia, schizophreniform, schizoaffective illness, PTSD, or conduct disorder.
3. T-score greater than/equal to 60 on baseline Social Responsiveness Scale
4. Meets criteria for substance use disorder in the three months prior to baseline.
5. Full scale intelligence < 70.
6. The symptoms are due to the direct physiological effects of drug abuse, or to a general medical or neurological condition.
7. Currently pregnant or lactating, or sexually active without using an acceptable method of contraception.
8. Failed an adequate trials (defined as four weeks of consecutive treatment at the minimally effective dose) or severe ill effects while on therapeutic doses of SSRI therapy.
9. Hypersensitivity or severe adverse reaction to methylphenidate.
10. History of fainting after exercise, syncope, a young family with sudden cardiac death, or known structural heart defect.
11. A serious history of adverse reactions (psychosis, severely increased activation compared to baseline) to methylphenidate or amphetamines.
12. Any chronic medical condition that requires medication that is contraindicated with SSRI or stimulant therapy, or any serious chronic or unstable medical disorder.
13. Medical contraindication to treatment with SSRI or stimulant therapy. -

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2013-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James J McGough, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At completion of open lisdexamfetamine, participants who achieved Clinical Global Impression Severity (CGI-S) SMD score < 4 were deemed sufficiently improved, and not randomized to adjunctive treatment. N=4 participants were sufficiently improved and completed study participation at study week 4, prior to randomization
Groups:
- Fluoxetine: All participants initially enrolled in open lisdexamfetamine treatment, followed by randomization to adjunctive fluoxetine at study week 4 and continuing to study week 12.
- Placebo: All participants initially enrolled in open lisdexamfetamine treatment, followed by randomization to adjunctive placebo at study week 4 and continuing through study week 12.
- Open Lisdexamfetamine: All eligible participants initially titrated to optimal dose open lisdexamfetamine beginning at baseline (week 0) and continuing to the end of study week 4.
Period: Open Lisdexamfetamine Titration
Arm/Group | Fluoxetine | Placebo | Open Lisdexamfetamine
Started | 0 | 0 | 34
Completed | 0 | 0 | 30
Not Completed | 0 | 0 | 4
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 3
Period: Double Blind Adjunctive Treatment
Arm/Group | Fluoxetine | Placebo | Open Lisdexamfetamine
Started | 12 (Adjunctive fluoxetine treatment was initiated at beginning of Period 2, at study week 4.) | 14 (Adjunctive placebo was initiated at beginning of Period 2, at study week 4.) | 0 (No one remained on lisdexamfetamine alone in Period 2.)
Completed | 10 | 11 | 0
Not Completed | 2 | 3 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: See Participant Flow descriptions.
Groups:
- Open Lisdexamfetamine: All eligible participants initially titrated to optimal dose open lisdexamfetamine from baseline through week 3.
- Fluoxetine: Randomized participants who competed open-label lisdexamfetamine titration from baseline through week 3, who continued to meet eligibility criteria, and then proceeded to adjunctive fluoxetine therapy from week 4 through week 12.
- Placebo: Randomized participants who competed open-label lisdexamfetamine titration from baseline through week 3, who continued to meet eligibility criteria, and then proceeded to adjunctive placebo from week 4 through week 12.
- Total: Total of all reporting groups
Arm/Group | Open Lisdexamfetamine | Fluoxetine | Placebo | Total
Number analyzed (Participants) | 34 | 12 | 14 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] — Columns for baseline measures are not additive, as fluoxetine and placebo groups are a subset of the original 34 participants entered into phase 1.
  years | 10.24 (2.58) | 9.97 (2.30) | 10.22 (2.74) | NA (NA) — Columns are not additive, as described above.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 5 | 5 | 23
  Male | 21 | 7 | 9 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 0 | 11
  Not Hispanic or Latino | 28 | 7 | 14 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 27 | 8 | 13 | 48
  More than one race | 5 | 4 | 1 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Wechsler Abbreviated Scale of Intelligence [Mean (Standard Deviation); unit: units on a scale] — Standard IQ measure for youth, frequently used in clinical studies, based on an administered test, with mean population score = 100.
  units on a scale | 103.16 (14.30) | 105.58 (15.56) | 101.69 (14.34) | NA (NA) — Columns not additive as described above.
Clinical Global Impression SMD Severity [Mean (Standard Deviation); unit: units on a scale] — A dimensional NIH measures used to quantify severity of severe mood dysregulation. Minimum score = 1. Maximum score = 7. Higher scores mean greater impairment.
  units on a scale | 4.82 (.52) | 4.75 (.46) | 4.83 (.72) | NA (NA) — Columns not additive as described above.
Affective Reactivity Index Parent Report [Mean (Standard Deviation); unit: units on a scale] — A parent completed dimensional measure of irritability on a scale of 0 to 14, with 14 being most severe.
  units on a scale | 8.91 (2.47) | 10.00 (1.95) | 8.57 (2.17) | NA (NA) — Columns not additive as described above.

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression-Severity-Severe Mood Dysregulation
Description: A dimensional clinician rating of overall SMD related impairment, modified by the National Institute of Mental Health to assess specific domains pertinent to Severe Mood Dysregulation. Minimum score = 1. Maximum score = 7. Higher scores means greater impairment.
Time Frame: Baseline through week 12.
Population: Compares groups lisdexamfetamine plus fluoxetine vs. lisdexamfetamine plus placebo over 12 week trial. Some participants discontinued as trial progressed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Fluoxetine: All participants initially enrolled in open lisdexamfetamine treatment, followed by randomization to adjunctive fluoxetine at week 4 continuing to week 12.
- Placebo: All participants initially enrolled in open lisdexamfetamine treatment, followed by randomization to adjunctive placebo at week 4 continuing through week 12.
- Open Lisdexamfetamine: All eligible participants initially titrated to optimal dose open lisdexamfetamine starting at baseline (week 0) and continuing through study week.
Arm/Group | Fluoxetine | Placebo | Open Lisdexamfetamine
Number analyzed (Participants) | 12 | 14 | 34
units on a scale
  Baseline | 4.91 (.53) | 3.62 (.48) | 4.30 (.32)
  Week 4: number analyzed (Participants) | 12 | 14 | 30
  Week 4 | 4.42 (.34) | 4.57 (.31) | 4.31 (.19)
  Week 5: number analyzed (Participants) | 12 | 14 | 0
  Week 5 | 4.15 (.36) | 3.51 (.32) |
  Week 6: number analyzed (Participants) | 12 | 14 | 0
  Week 6 | 3.67 (.34) | 3.90 (.33) |
  Week 7: number analyzed (Participants) | 10 | 14 | 0
  Week 7 | 3.61 (.37) | 3.59 (.34) |
  Week 8: number analyzed (Participants) | 10 | 13 | 0
  Week 8 | 3.42 (.39) | 3.37 (.34) |
  Week 10: number analyzed (Participants) | 10 | 11 | 0
  Week 10 | 3.45 (.42) | 3.11 (.35) |
  Week 12: number analyzed (Participants) | 10 | 11 | 0
  Week 12 | 3.51 (.38) | 3.30 (.36) |
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .58, Mixed Models Analysis — Group: F=.31, df=1/140; Partial linear regression using mixed model, assessing outcome variable over time (baseline to study week 12) and time2 (study weeks 4-12)
Statistical Analysis 2: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .85, Mixed Models Analysis — Partial linear regression using mixed model, assessing outcome variable over time (baseline to study week 12) and time2 (study weeks 4-12); Time: F=.03, df=1/140
Statistical Analysis 3: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .26, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Time2: F=1.28, df=1/140

2. Secondary Outcome: ADHD-IV Rating Scale
Description: A dimensional rating of ADHD symptoms, with scores ranging from 0 - 54, and higher scores indicating greater symptom severity.
Time Frame: Baseline through week 12.
Population: Participants discontinued as trial progressed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Fluoxetine: All participants initially enrolled in open lisdexamfetamine treatment, followed by randomization to adjunctive fluoxetine at end of study week 4 6 continuing through week 12.
- Placebo: All participants initially enrolled in open lisdexamfetamine treatment, followed by randomization to adjunctive placebo at end of study week 4 and continuing through week.
- Open Lisdexamfetamine: All eligible participants initially titrated to optimal dose open lisdexamfetamine at study visits 2-6.
Arm/Group | Fluoxetine | Placebo | Open Lisdexamfetamine
Number analyzed (Participants) | 12 | 14 | 34
units on a scale
  Baseline | 34.50 (1.97) | 34.31 (1.87) | 34.20 (1.15)
  Week 4: number analyzed (Participants) | 12 | 14 | 30
  Week 4 | 14.92 (1.97) | 18.64 (1.82) | 16.59 (1.21)
  Week 12: number analyzed (Participants) | 10 | 11 | 0
  Week 12 | 16.29 (2.10) | 11.93 (1.99) |
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .97, Mixed Models Analysis — Group: F=0.00, df=1/44; Partial linear regression using mixed model, assessing outcome variable over time (baseline through week 12) and time2 (weeks 4-12)
Statistical Analysis 2: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p < .0002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Time: F=136.22, df=1/44
Statistical Analysis 3: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p < .0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Time2: F=64.90, df=1/44

3. Secondary Outcome: Conners Parent Global Index
Description: Parent completed dimensional measure of ADHD symptoms, with score range from 0 - 30 and higher scores indicating more severe symptoms.
Time Frame: Baseline through week 3.
Population: Participants were assessed on this measure only during the Open Lisdexamfetamine phase. Some participant discontinued as trial progressed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Fluoxetine: All participants initially enrolled in open lisdexamfetamine treatment, followed by randomization to adjunctive fluoxetine at week 4 continuing tp week 12.
- Placebo: All participants initially enrolled in open lisdexamfetamine treatment, followed by randomization to adjunctive placebo at week 4 and continuing through week 12.
- Open Lisdexamfetamine: All eligible participants initially titrated to optimal dose open lisdexamfetamine beginning at baseline (week 0) and continuing through study week 4.
Arm/Group | Fluoxetine | Placebo | Open Lisdexamfetamine
Number analyzed (Participants) | 0 | 0 | 34
units on a scale
  Baseline |  |  | 15.91 (.82)
  Week 1: number analyzed (Participants) | 0 | 0 | 33
  Week 1 |  |  | 9.54 (.82)
  Week 2: number analyzed (Participants) | 0 | 0 | 33
  Week 2 |  |  | 10.60 (.85)
  Week 3: number analyzed (Participants) | 0 | 0 | 31
  Week 3 |  |  | 8.60 (.87)
Statistical Analysis 1: Comparison: Open Lisdexamfetamine; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Time: F=41.85, df=1/89, p<.0001; Linear regression of outcome change over time within single group

4. Secondary Outcome: Conners Global Index Emotional Lability Subscale - Parent Report
Description: A sub scale of the Conners Global Index, with scores ranging from 0 - 12, with higher scores indicating more impairment.
Time Frame: Baseline to week 3.
Population: Participants were assessed on this measure only during the Open Lisdexamfetamine phase. Some participants discontinues as trial progressed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Open Lisdexamfetamine: All eligible participants initially titrated to optimal dose open lisdexamfetamine beginning at baseline (week 0) and continuing through week 4.
Arm/Group | Fluoxetine | Placebo | Open Lisdexamfetamine
Number analyzed (Participants) | 0 | 0 | 34
units on a scale
  Baseline |  |  | 8.81 (.52)
  Week 1: number analyzed (Participants) | 0 | 0 | 33
  Week 1 |  |  | 5.90 (.52)
  Week 2: number analyzed (Participants) | 0 | 0 | 33
  Week 2 |  |  | 6.33 (.53)
  Week 3: number analyzed (Participants) | 0 | 0 | 31
  Week 3 |  |  | 5.45 (.55)
Statistical Analysis 1: Comparison: Open Lisdexamfetamine; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Time: F=26.65, df=1/92, p <.0001; Linear regression of outcome change over time within single group

5. Secondary Outcome: Conners Global Index Restless-Impulsive Subscale Parent Report
Description: A dimensional parent report measure of restless-impulsive symptoms, with scores ranging from 0 to 21, and higher scores indicating greater impairment.
Time Frame: Baseline through week 3.
Population: Participants were assessed on this measure only during the Open Lisdexamfetamine phase. Some participants discontinued as trial progressed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: All participants initially enrolled in open lisdexamfetamine treatment, followed by randomization to adjunctive placebo at week 4 though week 12.
Arm/Group | Fluoxetine | Placebo | Open Lisdexamfetamine
Number analyzed (Participants) | 0 | 0 | 34
units on a scale
  Baseline |  |  | 15.91 (.82)
  Week 1: number analyzed (Participants) | 0 | 0 | 33
  Week 1 |  |  | 9.55 (.82)
  Week 2: number analyzed (Participants) | 0 | 0 | 33
  Week 2 |  |  | 10.60 (.85)
  Week 3: number analyzed (Participants) | 0 | 0 | 31
  Week 3 |  |  | 8.60 (.87)
Statistical Analysis 1: Comparison: Open Lisdexamfetamine; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Time: F=40.35, df=1/89, p < .0001; Linear regression of outcome change over time within single group

6. Secondary Outcome: Conners Teacher Global Index
Description: Teacher completed dimensional measure of ADHD symptoms, with scores ranging from 0 - 30, and higher scores indicating more severe impairment.
Time Frame: Baseline through week 3.
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fluoxetine | Placebo | Open Lisdexamfetamine
Number analyzed (Participants) | 0 | 0 | 34
units on a scale
  Baseline |  |  | 18.13 (1.87)
  Week 1: number analyzed (Participants) | 0 | 0 | 33
  Week 1 |  |  | 13.21 (1.87)
  Week 2: number analyzed (Participants) | 0 | 0 | 33
  Week 2 |  |  | 10.18 (1.93)
  Week 3: number analyzed (Participants) | 0 | 0 | 31
  Week 3 |  |  | 8.31 (1.61)
Statistical Analysis 1: Comparison: Open Lisdexamfetamine; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Time: F=26.36, df=1/29, p <.0001; Linear regression of outcome change over time within single group

7. Secondary Outcome: Affective Reactivity Index - Parent Report
Description: A parent completed dimensional measure of emotional reactivity, with scores ranging from 0-12, and higher scores indicating greater severity.
Time Frame: Baseline through week 12.
Population: Some participants discontinued as trial progressed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fluoxetine | Placebo | Open Lisdexamfetamine
Number analyzed (Participants) | 12 | 14 | 34
units on a scale
  Baseline | 10.00 (.96) | 8.57 (.88) | 9.29 (.92)
  Week 4: number analyzed (Participants) | 12 | 14 | 30
  Week 4 | 7.58 (.96) | 7.71 (.88) | 6.87 (.59)
  Week 5: number analyzed (Participants) | 12 | 14 | 0
  Week 5 | 6.58 (.96) | 6.21 (.88) |
  Week 6: number analyzed (Participants) | 12 | 14 | 0
  Week 6 | 6.42 (.96) | 5.32 (.90) |
  Week 7: number analyzed (Participants) | 10 | 14 | 0
  Week 7 | 6.69 (1.00) | 6.49 (1.00) |
  Week 8: number analyzed (Participants) | 10 | 13 | 0
  Week 8 | 6.49 (1.00) | 5.62 (.90) |
  Week 10: number analyzed (Participants) | 10 | 11 | 0
  Week 10 | 6.74 (1.07) | 4.89 (.97) |
  Week 12: number analyzed (Participants) | 10 | 11 | 0
  Week 12 | 6.39 (1.00) | 5.30 (.94) |
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .44, Mixed Models Analysis — Group: F=.60, df=1/157; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p < .0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Time: F=22.39, df=1/157
Statistical Analysis 3: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .04, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Time2: F=4.40, df=1/157

8. Secondary Outcome: Revised Modified Overt Aggression Scale - Total Score
Description: A parent rated retrospective dimensional assessment of oppositional and aggressive behaviors, with scores ranging from 0-40, and higher scores indicating greater severity.
Time Frame: Baseline through week 12.
Population: Some participants discontinued as trial progressed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fluoxetine | Placebo | Open Lisdexamfetamine
Number analyzed (Participants) | 12 | 14 | 34
units on a scale
  Baseline | 22.23 (4.44) | 33.68 (4.08) | 26.03 (2.61)
  Week 4: number analyzed (Participants) | 12 | 14 | 30
  Week 4 | 14.44 (4.30) | 25.35 (3.98) | 17.93 (2.67)
  Week 5: number analyzed (Participants) | 12 | 14 | 0
  Week 5 | 13.72 (4.31) | 20.60 (4.19) |
  Week 6: number analyzed (Participants) | 12 | 14 | 0
  Week 6 | 10.00 (4.20) | 20.55 (3.98) |
  Week 7: number analyzed (Participants) | 10 | 14 | 0
  Week 7 | 13.19 (4.45) | 21.89 (4.32) |
  Week 8: number analyzed (Participants) | 10 | 13 | 0
  Week 8 | 14.09 (4.45) | 21.33 (4.08) |
  Week 10: number analyzed (Participants) | 10 | 11 | 0
  Week 10 | 12.61 (4.60) | 17.68 (4.47) |
  Week 12: number analyzed (Participants) | 10 | 11 | 0
  Week 12 | 14.29 (4.45) | 18.34 (4.32) |
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .05, Mixed Models Analysis — Group: F=3.81, df=1/145; [statistical method as in outcome 1, analysis 1]; No significant group*time interactions. Group trend likely due to baseline differences
Statistical Analysis 2: Comparison: Fluoxetine; Test type: Superiority; p = .0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Tie: F=15.28, df=1/145
Statistical Analysis 3: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .02, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Time2: F=5.42, df=1/145

9. Secondary Outcome: Clinical Global Impression - Improvement
Description: Percentage improved by treatment group
Time Frame: Percentage improved at week 4 for Open Lisdexamfetamine group and at week 12 for fluoxetine and placebo groups.
Population: Some participants discontinued as trial progressed.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluoxetine | Placebo | Open Lisdexamfetamine
Number analyzed (Participants) | 10 | 11 | 34
Participants | 7 | 7 | 8
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .76, Chi-squared; Chi Square = .10, df=1, p=.76

10. Secondary Outcome: Height
Description: A dimensional measure assessed in cms.
Time Frame: Baseline through week 12.
Population: Participants discontinued as trial progressed.
Measure: Least Squares Mean (Standard Error); unit: cm.
Arm/Group | Fluoxetine | Placebo | Open Lisdexamfetamine
Number analyzed (Participants) | 12 | 14 | 34
cm.
  Baseline | 140.25 (3.82) | 144.63 (3.53) | 142.37 (2.12)
  Week 1: number analyzed (Participants) | 12 | 14 | 32
  Week 1 | 140.05 (3.81) | 144.76 (3.53) | 142.35 (2.12)
  Week 2: number analyzed (Participants) | 12 | 14 | 32
  Week 2 | 139.95 (3.82) | 144.81 (3.53) | 142.43 (2.12)
  Week 3: number analyzed (Participants) | 12 | 14 | 30
  Week 3 | 140.26 (3.82) | 144.88 (3.53) | 142.59 (2.12)
  Week 4: number analyzed (Participants) | 12 | 14 | 30
  Week 4 | 140.56 (3.82) | 144.54 (3.53) | 142.59 (2.12)
  Week 5: number analyzed (Participants) | 12 | 14 | 0
  Week 5 | 140.11 (3.82) | 144.82 (3.53) |
  Week 6: number analyzed (Participants) | 12 | 14 | 0
  Week 6 | 140.21 (3.82) | 145.44 (3.53) |
  Week 7: number analyzed (Participants) | 10 | 14 | 0
  Week 7 | 140.55 (3.82) | 145.14 (3.53) |
  Week 8: number analyzed (Participants) | 10 | 13 | 0
  Week 8 | 140.81 (3.82) | 144.98 (3.53) |
  Week 10: number analyzed (Participants) | 10 | 11 | 0
  Week 10 | 140.83 (3.82) | 145.30 (3.54) |
  Week 12: number analyzed (Participants) | 10 | 11 | 0
  Week 12 | 140.98 (3.82) | 145.60 (3.53) |
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .38, Mixed Models Analysis — Group: F=.78, df=1/220; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .42, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Time: F=.66, df=1/220
Statistical Analysis 3: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .13, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Time2: F=.66, df=1/220

11. Secondary Outcome: Weight
Description: Weight in kg.
Time Frame: Baseline through week 12.
Population: Some participants discontinued as trial progressed.
Measure: Least Squares Mean (Standard Error); unit: kg.
Arm/Group | Fluoxetine | Placebo | Open Lisdexamfetamine
Number analyzed (Participants) | 12 | 14 | 34
kg.
  Baseline | 37.96 (5.26) | 47.26 (4.87) | 42.59 (3.16)
  Week 1: number analyzed (Participants) | 12 | 14 | 32
  Week 1 | 37.29 (5.26) | 46.39 (4.87) | 41.83 (3.16)
  Week 2: number analyzed (Participants) | 12 | 14 | 32
  Week 2 | 36.96 (5.26) | 45.56 (4.87) | 41.29 (3.16)
  Week 3: number analyzed (Participants) | 12 | 14 | 30
  Week 3 | 36.55 (5.26) | 45.06 (4.87) | 40.73 (3.16)
  Week 4: number analyzed (Participants) | 12 | 14 | 30
  Week 4 | 36.20 (5.26) | 45.22 (4.87) | 40.67 (3.16)
  Week 5: number analyzed (Participants) | 12 | 14 | 0
  Week 5 | 36.08 (5.26) | 44.80 (4.87) |
  Week 6: number analyzed (Participants) | 12 | 14 | 0
  Week 6 | 35.73 (5.26) | 44.34 (4.87) |
  Week 7: number analyzed (Participants) | 10 | 14 | 0
  Week 7 | 35.30 (5.26) | 44.72 (4.87) |
  Week 8: number analyzed (Participants) | 10 | 13 | 0
  Week 8 | 35.08 (5.26) | 44.08 (4.87) |
  Week 10: number analyzed (Participants) | 10 | 11 | 0
  Week 10 | 34.61 (5.26) | 44.16 (4.87) |
  Week 12: number analyzed (Participants) | 10 | 11 | 0
  Week 12 | 34.73 (5.26) | 43.05 (4.87) |
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .21, Mixed Models Analysis — Group: F=1.56, df=1/222; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p < .0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Time: F=63.11, df=1/222
Statistical Analysis 3: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .0004, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Time2: F=12.86, df=1/222

12. Secondary Outcome: Pulse
Description: Heart rate in beats per minute.
Time Frame: Baseline through week 12.
Population: Some participants discontinued as trial progressed.
Measure: Least Squares Mean (Standard Error); unit: beats per minute.
Arm/Group | Fluoxetine | Placebo | Open Lisdexamfetamine
Number analyzed (Participants) | 12 | 14 | 34
beats per minute.
  Baseline | 82.28 (3.26) | 84.64 (3.22) | 80.84 (2.30)
  Week 1: number analyzed (Participants) | 12 | 14 | 32
  Week 1 | 95.08 (3.16) | 85.21 (2.91) | 88.15 (2.13)
  Week 2: number analyzed (Participants) | 12 | 14 | 32
  Week 2 | 88.25 (3.15) | 81.64 (2.91) | 84.33 (2.13)
  Week 3: number analyzed (Participants) | 12 | 14 | 30
  Week 3 | 96.32 (3.26) | 85.79 (3.01) | 90.71 (2.26)
  Week 4: number analyzed (Participants) | 12 | 14 | 30
  Week 4 | 93.08 (3.15) | 83.21 (2.91) | 88.45 (2.23)
  Week 5: number analyzed (Participants) | 12 | 14 | 0
  Week 5 | 94.16 (3.26) | 83.00 (3.23) |
  Week 6: number analyzed (Participants) | 12 | 14 | 0
  Week 6 | 87.33 (3.15) | 90.55 (3.12) |
  Week 7: number analyzed (Participants) | 10 | 14 | 0
  Week 7 | 91.94 (3.55) | 90.00 (3.22) |
  Week 8: number analyzed (Participants) | 10 | 13 | 0
  Week 8 | 87.17 (3.40) | 85.10 (3.00) |
  Week 10: number analyzed (Participants) | 10 | 11 | 0
  Week 10 | 95.83 (3.55) | 82.90 (3.52) |
  Week 12: number analyzed (Participants) | 10 | 11 | 0
  Week 12 | 92.75 (3.55) | 90.62 (3.23) |
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .02, Mixed Models Analysis — Group: F=5.42, df=1/223; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .18, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Time: F=1.77, df=1/223
Statistical Analysis 3: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .49, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Time2: F=.47, df=1/223

13. Secondary Outcome: Systolic Blood Pressure
Description: Systolic Blood Pressure measured in mmHG
Time Frame: Baseline through week 12.
Population: Some participants discontinued as trial progressed.
Measure: Least Squares Mean (Standard Error); unit: mm Hg.
Arm/Group | Fluoxetine | Placebo | Open Lisdexamfetamine
Number analyzed (Participants) | 12 | 14 | 34
mm Hg.
  Baseline | 107.85 (4.01) | 106.68 (3.92) | 107.40 (2.69)
  Week 1: number analyzed (Participants) | 12 | 14 | 32
  Week 1 | 99.42 (3.89) | 111.71 (3.60) | 106.03 (2.53)
  Week 2: number analyzed (Participants) | 12 | 14 | 32
  Week 2 | 104.83 (3.89) | 110.36 (3.60) | 107.48 (2.53)
  Week 3: number analyzed (Participants) | 12 | 14 | 30
  Week 3 | 109.20 (4.01) | 109.89 (3.70) | 110.73 (2.67)
  Week 4: number analyzed (Participants) | 12 | 14 | 30
  Week 4 | 112.00 (3.89) | 110.07 (3.60) | 111.77 (2.65)
  Week 5: number analyzed (Participants) | 12 | 14 | 0
  Week 5 | 109.57 (4.01) | 104.20 (3.93) |
  Week 6: number analyzed (Participants) | 12 | 14 | 0
  Week 6 | 111.58 (3.89) | 108.98 (3.80) |
  Week 7: number analyzed (Participants) | 10 | 14 | 0
  Week 7 | 112.04 (4.31) | 112.80 (3.92) |
  Week 8: number analyzed (Participants) | 10 | 13 | 0
  Week 8 | 111.20 (4.31) | 110.94 (3.96) |
  Week 10: number analyzed (Participants) | 10 | 11 | 0
  Week 10 | 112.25 (4.31) | 105.67 (4.23) |
  Week 12: number analyzed (Participants) | 10 | 11 | 0
  Week 12 | 116.15 (4.31) | 113.90 (3.93) |
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .90, Mixed Models Analysis — Group: F=.02, df=1/223; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .21, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Time: F=1.60, df=1/223
Statistical Analysis 3: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .73, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Time2: F=.12, df=1/223

14. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic Blood pressure measured in mmHG.
Time Frame: Baseline through week 12.
Population: Some participants discontinued as trial progressed.
Measure: Least Squares Mean (Standard Error); unit: mm Hg.
Arm/Group | Fluoxetine | Placebo | Open Lisdexamfetamine
Number analyzed (Participants) | 12 | 14 | 34
mm Hg.
  Baseline | 68.86 (2.36) | 66.40 (2.34) | 67.39 (1.56)
  Week 1: number analyzed (Participants) | 12 | 14 | 32
  Week 1 | 71.33 (2.27) | 69.50 (2.10) | 69.15 (1.45)
  Week 2: number analyzed (Participants) | 12 | 14 | 32
  Week 2 | 66.00 (2.27) | 66.79 (2.10) | 66.63 (1.45)
  Week 3: number analyzed (Participants) | 12 | 14 | 30
  Week 3 | 68.74 (2.36) | 62.82 (2.18) | 67.21 (1.56)
  Week 4: number analyzed (Participants) | 12 | 14 | 30
  Week 4 | 71.17 (2.27) | 66.21 (2.10) | 69.31 (1.53)
  Week 5: number analyzed (Participants) | 12 | 14 | 0
  Week 5 | 71.17 (2.36) | 65.17 (2.34) |
  Week 6: number analyzed (Participants) | 12 | 14 | 0
  Week 6 | 69.58 (2.27) | 70.61 (2.25) |
  Week 7: number analyzed (Participants) | 10 | 14 | 0
  Week 7 | 68.14 (2.58) | 70.64 (2.34) |
  Week 8: number analyzed (Participants) | 10 | 13 | 0
  Week 8 | 68.06 (2.46) | 68.40 (2.17) |
  Week 10: number analyzed (Participants) | 10 | 11 | 0
  Week 10 | 70.81 (2.58) | 67.06 (2.56) |
  Week 12: number analyzed (Participants) | 10 | 11 | 0
  Week 12 | 77.11 (2.58) | 70.05 (2.34) |
Statistical Analysis 1: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .15, Mixed Models Analysis — Group: F=2.05, df=1/223; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .59, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Time: F=.29, df=1/223
Statistical Analysis 3: Comparison: Fluoxetine vs Placebo; Test type: Superiority; p = .14, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Time2: F=2.15, df=1/223

15. Other Pre Specified Outcome: Pediatric Anxiety Rating Scale
Description: Clinician completed dimensional assessment of anxiety symptoms.
Time Frame: Baseline through week 12.
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Children's Depression Rating Scale
Description: Clinician completed dimensional rating of depressive symptoms.
Time Frame: Baseline through week 12.
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Affective Reactivity Index Child Report
Description: Dimensional self-report of irritability, with total score 1-12, and higher scores indicating greater severity.
Time Frame: Baseline through week 12.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline through study week 12.
Description: Adverse events were collected via structured ratings, including the Columbia Suicide Severity Rating Scale and the Side Effects Rating Scale.
Groups:
- Fluoxetine: All participants initially enrolled in open lisdexamfetamine treatment, followed by randomization to adjunctive fluoxetine at week 4 and continuing though week 12.
- Placebo: All participants initially enrolled in open lisdexamfetamine treatment, followed by randomization to adjunctive placebo at study week 4 and continuing through week 12.
- Open Lisdexamfetamine: All eligible participants initially titrated to optimal dose open lisdexamfetamine from baseline through week 4.
Arm/Group | Fluoxetine | Placebo | Open Lisdexamfetamine
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14 | 0/34
Other Adverse Events (participants affected / at risk) | 8/12 | 10/14 | 30/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoxetine (N=12) | Placebo (N=14) | Open Lisdexamfetamine (N=34)
Wish to be dead (Psychiatric disorders) | 1 (3) | 2 (2) | 0 (0) — Endorsed on Columbia Suicide Severity Rating Scale
Suicidal ideation without intent (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Endorsed on Columbia Suicide Severity Rating Scale
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 5 (8) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Feeling drowsy/sleep (General disorders) | 1 (2) | 1 (1) | 4 (5) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Dry mouth (General disorders) | 0 (0) | 3 (3) | 4 (6) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Stomach pain/ache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (5) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Nausea/vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Frequent urination (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Restless/uncomfortable urge to move (General disorders) | 1 (1) | 2 (4) | 1 (2) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Heart skips beats (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Racing heart (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Trouble sleeping (Psychiatric disorders) | 1 (1) | 4 (6) | 9 (15) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Sleeplessness (Psychiatric disorders) | 1 (6) | 2 (4) | 4 (9) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Nightmares (Psychiatric disorders) | 0 (0) | 2 (3) | 1 (1) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Excessive sweating (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Tremor/shakiness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Decreased appetite (General disorders) | 7 (24) | 6 (11) | 21 (51) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Tics (Nervous system disorders) | 2 (2) | 3 (3) | 4 (7) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Euphoria (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Talks less with others (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Bites fingernails (Nervous system disorders) | 3 (5) | 2 (6) | 5 (7) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.
Prone to crying (Psychiatric disorders) | 0 (0) | 3 (3) | 6 (9) — Clinically significant symptom with post baseline onset based on parent completed Physical Symptoms Checklist.

LIMITATIONS AND CAVEATS:
Study was designed as an initial feasibility and proof of concept trial. Initial power analysis suggested need to randomize N=50 participants. Recruitment was much more difficult than expected, leading to small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No